CLINICAL TRIAL: NCT02447510
Title: Crevicular Fluid Growth Factors Release Profile Following the Use of Platelets Rich Fibrin (PRF) and Plasma Rich Growth Factors (PRGF) in Treating Periodontal Intrabony Defects (Randomized Clinical Trial)
Brief Title: Growth Factors Release of PRF and PRGF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Y Gamal, professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ain Shams Universty
Record Dates: First submitted 2015-05-06; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- group 1 (Other): bone substitute grafting material applied to the defect site control (n=10)
  Interventions: Procedure: group 1 bio-oss bone xenograft
- group 2 (Other): experimental platelet rich growth factor PRGF applied to the defect site (n=10) G2
  Interventions: Procedure: group 2 platelet rich in growth factor (autogenous platelet rich in growth factor)
- group 3 (Other): platelet rich fibrin PRF applied to the defect site (n=10) G3.
  Interventions: Procedure: group 3 platelet rich fibrin (autogenous platelet rich fibrin)

INTERVENTIONS:
Procedure: group 1 bio-oss bone xenograft — bone substitute (bio-oss)
  Other Names: bio-oss bone xenograft
  Arms: group 1
Procedure: group 2 platelet rich in growth factor (autogenous platelet rich in growth factor) — platelet rich in growth factor (autogenous platelet rich in growth factor)
  Other Names: PRGF
  Arms: group 2
Procedure: group 3 platelet rich fibrin (autogenous platelet rich fibrin) — platelet rich fibrin (autogenous platelet rich fibrin)
  Other Names: PRF
  Arms: group 3

SUMMARY:
Background: platelet concentrate could enhance growth factors (GF) crevicular fluid levels which might be crucial to proper tissue repair and wound healing. However, the open usually contaminated nature of periodontal defects could affect negatively GF availability and activity. To test this assumption, this study was designed to evaluate levels of VEGF and PDGF-BB in gingival crevicular fluid (GCF) during the early stages of healing of localized intrabony defects treated with platelet rich in growth factor (PRGF) and platelet rich fibrin (PRF) as compared with xenograft defect filling control.

Methods: Thirty non-smoking patients with severe chronic periodontitis participated in this prospective, randomized and single blinded trial. Each patient contributed one interproximal defect that was randomly assigned to the bone substitute grafting control (n=10) G1, experimental PRGF (n=10) G2 and PRF (n=10) G3. Plaque index, gingival index, probing depth (PD), clinical attachment level (CAL) and the intrabony depth of the defect (IBD) were measured at baseline for patient enrollment. Gingival crevicular fluid (GCF) samples were collected on days 1 and 3, 7, 14, 21, and 30 days after therapy. The primary outcome variable was the change in VEGF and PDGF-BB levels for sites treated by PRGF and PRF compared to that of the xenograft treated cases.

DETAILED DESCRIPTION:
Owing to the lots of challenges that facing the use of recombinant growth factors in periodontal therapy, it is important to look for an alternative that combine ease of preparation and physiologic mode of delivery. Platelet concentrate has been developed for this purpose with many debates about the duration of GF availability in the defect area. Platelet-rich fibrin (PRF) is a leucocyte- and platelet-rich fibrin biomaterial. This dense fibrin membrane was claimed to releases high quantities of three main growth factors (Transforming Growth Factor b-1 (TGFβ-1), platelet derived growth factor AB, PDGF-AB; vascular endothelial growth factor, VEGF) and an important coagulation matricellular glycoprotein (thrombospondin-1, TSP-1). It has a natural fibrin framework that can protect growth factors from proteolysis. It is shown that PRF can release growth factors gradually and keep their activity to a relatively long period compared with platelet rich plasma (PRP). Levels of released TGF-1 and PDGF-AB markedly increased and reached the highest amount at day , then decreased mildly. In contrast, PRP experienced uncontrollable and short-term release of TGF-1 and PDGF-AB, which reached the highest amount at day 1 and then decreased rapidly.Clinically, it was found that PRF can improve clinical parameters associated with human intrabony periodontal defects and BPBM (bovine porous bone mineral) has the ability to augment effects of PRF in reducing pocket depth, improving clinical attachments levels, and promoting defect fill. On the other hand studies reported similar PD (probing depth) reduction, CAL (clinical attachment level) gain, and bone fill at sites treated with PRF or PRP compared with conventional open flap debridement.

Preparation rich in growth factors (PRGF-Endoret) technology was claimed to circumvent many of the limitations of other reported platelet-rich preparations. Sodium citrate and calcium chloride are used as an anticoagulant and a clot activator, respectively. Addition of calcium chloride promotes the formation of native thrombin, mimicking the physiological clotting process and enabling a more sustained release of growth factors, which might be crucial to proper tissue repair and wound healing. Moreover, this procedure obviates immunological reactions and the risk of disease transmission associated with the use of exogenous bovine thrombin. Anitua et al reported that PRGF contains a moderately elevated platelet concentration of ~6x105 platelets, which has been reported to induce the optimal biological benefit. Lower platelet concentrations can lead to suboptimal effects, whereas higher concentrations might have an inhibitory effect. PRGF application after extraction improved the healing process in diabetic patients by accelerating socket closure (epithelialization) and tissue maturation, proving the association between PRGF use and improved wound healing in diabetic patients.

In the present study it was proposed that the opened, constantly contaminated nature periodontal defects could be a source of continuous catabolic bacterial and tissue enzymes and binding proteins that affect platelet concentrate contained GF availability and activity. To confirm this assumption, this study was designed to evaluate levels of platelet derived growth factor - BB (PDGF-BB) and vascular endothelial cell growth factor (VEGF) in GCF during the early stages of healing for sites treated with PRF and PRGF in intrabony periodontal defects and to correlate GF levels with the clinical findings. This could figure out the potentials of these 2 commonly used platelet concentrate in the periodontal defects ecology.

ELIGIBILITY:
Inclusion Criteria:

1. no systemic diseases which could influence platelet concentration or the outcome of therapy;
2. good compliance with plaque control instructions following initial therapy;
3. teeth involved were all vital with no mobility ;
4. each subject contributed a single predominately 2 or 3-wall intrabony interproximal defect around premolar or molar teeth without furcation involvement;
5. selected intrabony defects (IBDs) measured from the alveolar crest to the defect base in diagnostic periapical radiographs of ≥ 3 mm;
6. selected probing depth (PD) ≥ 6 mm and clinical attachment loss (CAL) ≥ 5 mm at the site of intraosseous defects four weeks following initial cause-related therapy;
7. availability for the follow-up and maintenance program;
8. absence of periodontal treatment during the previous year;
9. absence of systemic medications that could affect healing or antibiotic treatment during the previous 6 months; and
10. absence of occlusal interferences or open interproximal contacts (diastema, flaring or both).

Exclusion Criteria:

1. smokers and Pregnant females were excluded from participating in the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameters for the study were the crevicular fluid VEGF and PDGF-BB levels at 1 day | 1 day
crevicular fluid VEGF and PDGF-BB levels at 3day | 3 days
crevicular fluid VEGF and PDGF-BB levels at 7 day | 7 days
crevicular fluid VEGF and PDGF-BB levels at 14 day | 14 days
crevicular fluid VEGF and PDGF-BB levels at 21 day | 21 days
crevicular fluid VEGF and PDGF-BB levels at 30 day | 30 days

SECONDARY OUTCOMES:
Secondary efficacy parameters included pocker depth at 6 months after surgery. | 6 months
Secondary efficacy parameters included pocker depth at 9 months after surgery. | 9 months
Secondary efficacy parameters included radiographic intrabony defect depth measurements 9 months after surgery. | 9 months
Secondary efficacy parameters included clinical attachment level at 6 months after surgery. | 6 months
Secondary efficacy parameters included clinical attachment level at 9 months after surgery. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Y Gamal, PhD, Study Chair — Ain Shams Universty
Locations (1):
- Ain Shams Universty, Cairo, Nasr City, Egypt